CLINICAL TRIAL: NCT01896024
Title: Effects of Motive-Oriented Therapeutic Relationship in the Early-Phase Treatment of Borderline Personality Disorder
Acronym: MOTR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Ueli Kramer, PhD, University of Lausanne Hospitals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SNSF 100014-134562
Record Dates: First submitted 2013-07-05; First posted 2013-07-11 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Borderline Personality Disorder
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- General Psychiatric Management (GPM; Gunderson & Links, 2008) (Active Comparator): psychodynamic-psychiatric treatment for borderline personality disorder
  Interventions: Behavioral: Psychiatric Management
- GPM plus Motive-Oriented Therapeutic Relationship (Experimental): use of Plan Analysis and Motive-oriented therapeutic relationship, as add-on variable to GPM
  Interventions: Behavioral: Psychiatric Management; Behavioral: Motive-oriented therapeutic relationship/Plan Analysis

INTERVENTIONS:
Behavioral: Psychiatric Management
Behavioral: Motive-oriented therapeutic relationship/Plan Analysis
  Arms: GPM plus Motive-Oriented Therapeutic Relationship

SUMMARY:
The present research aims at examining the effectiveness of a specific set of therapist relational interventions and attitudes, called the Motive-Oriented Therapeutic Relationship (MOTR), based on Plan Analysis (Caspar, 2007) in the early-phase treatment of patients diagnosed with Borderline Personality Disorder.

The investigators intend to include N = 80 outpatients diagnosed with Borderline Personality Disorder, consulting at the Outpatient Personality Disorder Program of the Karl Jaspers Clinical Unit, in collaboration with the Institute of Psychotherapy, at the Department of Psychiatry-CHUV, University of Lausanne and in collaboration with the University of Berne, Switzerland. Patients are assigned by chance to two treatment conditions 1) Control condition (General Psychiatric Management; Gunderson & Links, 2008) and 2) MOTR-condition. The investigators hypothesize better results in the MOTR-condition, as compared to the control condition in terms of symptom reduction pre-post.

The conduct of the study represents a significant contribution to the understanding and enhancement of relationship aspects in the treatment of patients diagnosed with Borderline Personality Disorder which may be of potential benefit for these patients.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV Borderline Personality Disorder;
* between 18 and 65 yrs of age

Exclusion Criteria:

* DSM-IV psychotic disorders,
* mental retardation,
* substance abuse in the forefront

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2010-06; Primary Completion 2013-05 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Outcome Questionnaire -45.2 (Lambert et al., 2004) | 3 months
  pre- post- intervention in a randomized controlle trial; measure of symptom reduction over 3 months

SECONDARY OUTCOMES:
Inventory of Interpersonal Problems (Horowitz et al., 1988) | 3 months
  Measure of interpersonal problems after 3 months of therapy

OTHER OUTCOMES:
Borderline Symptom List (Bohus, 2009) | 3 months
  Symptom reduction of borderline symptoms over 3 months of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry-CHUV, University of Lausanne, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Result] Kramer U, Berger T, Kolly S, Marquet P, Preisig M, de Roten Y, Despland JN, Caspar F. Effects of motive-oriented therapeutic relationship in early-phase treatment of borderline personality disorder: a pilot study of a randomized trial. J Nerv Ment Dis. 2011 Apr;199(4):244-50. doi: 10.1097/NMD.0b013e3182125d19. PMID 21451348
- [Result] Kramer U, Kolly S, Berthoud L, Keller S, Preisig M, Caspar F, Berger T, de Roten Y, Marquet P, Despland JN. Effects of motive-oriented therapeutic relationship in a ten-session general psychiatric treatment of borderline personality disorder: a randomized controlled trial. Psychother Psychosom. 2014;83(3):176-86. doi: 10.1159/000358528. Epub 2014 Apr 17. PMID 24752034
- [Result] Kramer U, Fluckiger C, Kolly S, Caspar F, Marquet P, Despland JN, de Roten Y. Unpacking the effects of therapist responsiveness in borderline personality disorder: motive-oriented therapeutic relationship, patient in-session experience, and the therapeutic alliance. Psychother Psychosom. 2014;83(6):386-7. doi: 10.1159/000365400. Epub 2014 Oct 16. No abstract available. PMID 25324025
- [Derived] Sallin L, Geissbuehler I, Grandjean L, Beuchat H, Martin-Soelch C, Pascual-Leone A, Kramer U. Self-Contempt, the Working Alliance and Outcome in Treatments for Borderline Personality Disorder: An Exploratory Study. Psychother Res. 2021 Jul;31(6):765-777. doi: 10.1080/10503307.2020.1849848. Epub 2020 Nov 30. PMID 33256540
- [Derived] Storebo OJ, Stoffers-Winterling JM, Vollm BA, Kongerslev MT, Mattivi JT, Jorgensen MS, Faltinsen E, Todorovac A, Sales CP, Callesen HE, Lieb K, Simonsen E. Psychological therapies for people with borderline personality disorder. Cochrane Database Syst Rev. 2020 May 4;5(5):CD012955. doi: 10.1002/14651858.CD012955.pub2. PMID 32368793
- [Derived] Penzenstadler L, Kolly S, Rothen S, Khazaal Y, Kramer U. Effects of substance use disorder on treatment process and outcome in a ten-session psychiatric treatment for borderline personality disorder. Subst Abuse Treat Prev Policy. 2018 Feb 26;13(1):10. doi: 10.1186/s13011-018-0145-6. PMID 29482597